CLINICAL TRIAL: NCT02772016
Title: Therapeutic Effect of Colla Corii Asini on Improving Anemia and Hemoglobin Composition in Pregnant Women With Thalassemia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yanfang Li (Other)
Responsible Party: Sponsor-Investigator, Yanfang Li, Dr., The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine
Organization: The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TH-1
Record Dates: First submitted 2016-04-15; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-04

CONDITIONS: Thalassemia
MeSH Terms: conditions — Thalassemia | interventions — colla corii asini

ARMS (2):
- Intervention group (Experimental): Patients in the treatment group received daily 15 g oral Colla corii asini(Shandong Dong-E E-Jiao Co., Ltd) in powder form for 4 consecutive weeks. The dosage was adjusted to 10 g per day for 6 consecutive weeks if patients encounter any of the following side effects: swollen gums, dry or sore throat, ulcers in oral cavity.
  Interventions: Drug: Colla corii asini
- Control group (No Intervention): Patients in control groups do not receive any intervention.

INTERVENTIONS:
Drug: Colla corii asini — 15 g of Colla corii asini in powder form daily for 4 weeks
  Arms: Intervention group

SUMMARY:
Seventy-two pregnant patients diagnosed of minor or intermediate beta thalassemia with mild anemia were randomly assigned to treatment group and control group. Patients in the treatment group were given 15 g of Colla corii asini in powder form daily for 4 weeks while the control group were observed and followed up in the same period without any treatments. Levels of hemoglobin(Hb), serum iron (SI), serum ferritin (SF) and three types of hemoglobin components [adult hemoglobin (HbA), fetal hemoglobin (HbF), minor adult hemoglobin (HbA2)] were measured before and after treatments.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women diagnosed as thalassemia carriers by genetic test with clinical presentation of minor or intermediate β- thalassemia;
* patients with mild anemia (80 g/L≤ Hb<110 g/L) prior to study enrollment;
* singleton pregnancy;
* patients having not received blood transfusion or any forms of anti-anemia treatment in Western Medicine or Traditional Chinese Medicine in the last 12 weeks;
* informed consent obtained.

Exclusion Criteria:

* patients with severe thalassemia;
* patients with severe anemia (Hb<80 g/L) prior to study enrollment;
* twin or multiple pregnancies;
* patients with any of the following abnormalities: immunodeficiency, primary diseases involving cardiovascular system, liver, kidney, gastrointestinal tract, endocrine system and hematological system;
* allergic to two or more drugs;
* patients with mental illness or poor compliance to medical treatment;
* patients having received blood transfusion or any forms of anti-anemia treatment in Western medicine or Traditional Chinese Medicine in the last 12 weeks;
* no informed consent obtained.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin(Hb) | Four weeks
  the change of hemoglobin(g/L)
Adult hemoglobin(HbA) | Four weeks
  the change of adult hemoglobin(%)
Fetal hemoglobin(HbF) | Four weeks
  the change of fetal hemoglobin(%)
Minor adult hemoglobin(HbA2) | Four weeks
  the change of minor adult hemoglobin(%)

SECONDARY OUTCOMES:
Serum iron(SI) | Four weeks
  the change of serum iron (umol/L)
Serum ferritin(SF) | Four weeks
  the change of serum ferritin (ng/mL)
Adverse effect | Four weeks
  total white blood count(×109/L)
Adverse effect | Four weeks
  platelet count(×109/L)
Adverse effect | Four weeks
  percentage of neutrophil(%)
Adverse effect | Four weeks
  serum alanine aminotransferase(U/L)
Adverse effect | Four weeks
  serum aspartate aminotransferase(U/L)
Adverse effect | Four weeks
  urea nitrogen (mmol/L)
Adverse effect | Four weeks
  serum creatinine(umol/L)

CONTACTS AND LOCATIONS:
Locations (1):
- the first affiliated hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Voskaridou E, Balassopoulou A, Boutou E, Komninaka V, Christoulas D, Dimopoulou M, Delaki EE, Loukopoulos D, Terpos E. Pregnancy in beta-thalassemia intermedia: 20-year experience of a Greek thalassemia center. Eur J Haematol. 2014 Dec;93(6):492-9. doi: 10.1111/ejh.12387. Epub 2014 Jun 26. PMID 24889414
- [Background] Costa D, Capuano M, Sommese L, Napoli C. Impact of epigenetic mechanisms on therapeutic approaches of hemoglobinopathies. Blood Cells Mol Dis. 2015 Aug;55(2):95-100. doi: 10.1016/j.bcmd.2015.05.004. Epub 2015 May 12. PMID 26142322
- [Background] Pavord S, Myers B, Robinson S, Allard S, Strong J, Oppenheimer C; British Committee for Standards in Haematology. UK guidelines on the management of iron deficiency in pregnancy. Br J Haematol. 2012 Mar;156(5):588-600. doi: 10.1111/j.1365-2141.2011.09012.x. PMID 22512001